CLINICAL TRIAL: NCT01156519
Title: Detection of Infra-clinic Cortisol Adenoma (ACIC) in a Population of Android Obese With High Metabolic Risk: Contribution of Salivary Cortisol at 23 Hours
Brief Title: Contribution of Salivary Cortisol in the Detection of Infra-clinic Cortisol Adenoma (ACIC)
Acronym: ACIC
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Number of patients with a serum cortisol > 18 ng/ml reached
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 09/12-I
Record Dates: First submitted 2010-06-29; First posted 2010-07-05 (Estimated); Last update posted 2014-07-22 (Estimated); Status verified 2014-07

CONDITIONS: Obesity
Keywords: Infra-clinic cortisol adenoma; Salivary cortisol; Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Salivary cortisol (Other)
  Interventions: Other: Salivary Cortisol

INTERVENTIONS:
Other: Salivary Cortisol — * Day 1: 1st salivary cortisol at 23 hours
  * Day 2: 2nd salivary cortisol at 23 hours and administration of dexamethasone (for overnight 1-mg dexamethasone suppression test)
  * Day 3: serum cortisol at 8 am
  * Between Day 4 and Month 3: if serum cortisol at 8 am > 18ng/mL:
  * Cortisol for 24 hours
  * dexamethasone suppression test (2mg/j during 2 days)
  * Cortisol and ACTH cycle
  * Noriodocholesterol scintigraphy

SUMMARY:
The main objective of the study is to assess the sensitivity of the salivary cortisol dosage at 23 hours compared to the serum cortisol dosage at 8 am after overnight 1-mg dexamethasone suppression test (Suppression of serum cortisol <1.8 μg/dL ) as the reference method for the detection of ACIC in obese subjects

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years)
* Signed informed consent
* Subjects affiliated with an appropriate social security system
* Body mass index above 30 kg/m2 and
* Pathological waist circumference according to criteria of NCEP ATPIII (men : 94 cm and women : 80 cm)

Exclusion Criteria:

* Pregnancy
* Sepsis
* Recent surgery (less than 30 days)
* Any recent severe acute conditions requiring hospitalisation (less than 30 days)
* Recent use (< 7 days) of oral steroids, inhaled, dermal, collyrium, infiltration
* Long-term oral corticosteroids
* Nicotinic substitute or per os licorice in 2 weeks before the inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 514 (Actual)
Dates: Start 2010-06; Primary Completion 2013-12 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Number of patients with positive salivary cortisol dosage among patients with positive serum cortisol dosage
  The main objective of the study is to assess the sensitivity of the salivary cortisol dosage at 23 hours compared to the serum cortisol dosage at 8 am after overnight 1-mg dexamethasone suppression test as the reference method for the detection of ACIC in obese subjects

SECONDARY OUTCOMES:
Number of patients with negative salivary cortisol dosage among patients with negative serum cortisol dosage
  To evaluate specificity, negative predictive value, positive predictive value and diagnostic accuracy of salivary cortisol compared to serum cortisol at 8 am after overnight 1-mg dexamethasone suppression test
Comparing the results of salivary cortisol dosage and serum cortisol dosage
  To evaluate concordance between salivary cortisol dosage and serum cortisol dosage
Comparing the results of the two salivary samples
  To evaluate the concordance of the two salivary samples
Number of patients with metabolic complications of obesity among patients with ACIC
  To evaluate the link between ACIC and metabolic complications of obesity (insulin resistance, IFG, type 2 diabetes, NAFLD…)
Number of patients with severe type 2 diabetes among patients with ACIC
  To evaluate the relationship between ACIC and severity of type 2 diabetes, if established.

CONTACTS AND LOCATIONS:
Overall Officials: Bertrand CARIOU, Pr, Principal Investigator — Nantes University Hospital
Locations (1):
- Nantes University Hospital, Nantes, France